CLINICAL TRIAL: NCT02058056
Title: Early Prophylactic Cranial Irradiation With Hippocampal Avoidance in Patients With Limited Disease Small-cell Lung Cancer. A Multicenter Phase II Trial
Brief Title: Early Hippocampal Avoidance Prophylactic Cranial Irradiation in Patients With LD SCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 15/12
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Small-Cell Lung Cancer
Keywords: Early prophylactic; cranial irradiation; hippocampal avoidance; limited disease small-cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: HA-PCI treatment (Experimental): Irradiation HA-PCI concomitant to the second cycle of CHT and to tRT for patients with LD SCLC
  Interventions: Radiation: Irradiation: HA-PCI

INTERVENTIONS:
Radiation: Irradiation: HA-PCI — 25 Gy in 10 daily factions, five times a week

SUMMARY:
The main objective of this trial is to assess NCF after early HA-PCI concomitant to the second cycle of CHT and to tRT for patients with LD SCLC.

DETAILED DESCRIPTION:
About 15% of all lung cancers are small cell lung cancer (SCLC). SCLC is a high-grade, neuroendocrine carcinoma of the lung. Limited disease (LD) SCLC is confined to the hemithorax of origin, the mediastinum, or the supraclavicular nodes, which can be encompassed within a tolerable radiation therapy port. About 30% of all SCLC are LD at diagnosis. The median overall survival (OS) in LD SCLC is approximately 20 months, with an expected 5-year survival of less than 15%.

SCLC is characterized by rapid growth and early dissemination. The standard treatment of LD SCLC involves multimodality therapy with concurrent thoracic radiotherapy (tRT) and chemotherapy (CHT) with cisplatin and etoposide.

Recurrence in the brain is usually the primary site of treatment failure in SCLC and is associated with significant morbidity; and consequently often the cause of death. Occult early dissemination of SCLC has frequently occurred prior to the time of diagnosis. In patients with brain metastasis two randomized trials showed an overall 5-year rate of brain metastasis of 59% without prophylactic cranial irradiation (PCI) compared to 43% with PCI. However the rate of brain metastasis with PCI is still very high.

About 50% of patients with SCLC will develop brain metastases some time during the course of their disease. Therefore PCI is recommended in case of good response to CHT and tRT. PCI has shown to improve overall survival in patients with LD who have achieved a complete or partial remission after initial chemoradiotherapy. CHT might achieve insufficient drug levels in the brain. Therefore, an up-front PCI could treat occult brain metastases at a preclinical state and may increase the permeability of the blood-brain barrier for CHT products.

When evaluating PCI it is important to weigh the reduced incidence of brain metastases against the potential risk of deficits resulting from the treatment itself, including deteriorations in neurocognitive functions (NCF) or quality of life (QoL).

A possibility to reduce long-term neurocognitive effects due to PCI is the sparing of the hippocampus. Recent technological advancements in radiation oncology delivery enable the avoidance of the hippocampus. A PCI with hippocampus avoidance (HA-PCI) can reduce memory loss due to radiation.

Prospective neurocognitive testing has been increasingly used in trials for patients with CNS tumors and in patients with brain metastases in order to determine the risks versus benefits of different treatment approaches. For this trial, the choice for NCF assessments follows the recommendation provided by Meyers and Brown (2006). This neurocognitive battery for the use in multinational drug trials with neurocognitive endpoints consists of four standardized psychometric instruments, i.e. the Hopkins Verbal Learning Test, the Controlled Oral Word Association Test (COWAT) and the Trail Making Part A and Part B (TMT A/B). These tests have been shown to be sensitive to the neurotoxic effects of cancer treatment in clinical trials and cover several cognitive functions (memory, verbal fluency, visual-motor speed, executive function). In addition, published normative data are available that take into account age, and where appropriate, education and sex. To minimize the effects of repeated administration alternate forms can be used and test administration is highly standardized. The same battery of tests has been used in trials conducted by the Radiation Therapy Oncology Group (RTOG) (e.g. Wolfson 2011), and one or several of these three tests were applied in most of the studies mentioned above. Using the same tests across trials is important in order to be able to compare results of different trials. It has been shown that performing a cognitive test battery consisting of five cognitive tests (and a QoL assessment) in a multi-site trial and cooperative group setting (i.e. a RTOG trial) in patients with brain metastases is feasible.

NCF can be affected by a number of factors such as the volume of brain metastases, disease progression, other treatments (e.g. surgery, chemo- or endocrine therapy), medications and psychological factors such as anxiety and distress. These factors should be considered when evaluating the actual neurocognitive effect of concomitant CHT, tRT and PCI.

Rationale for performing the trial PCI is part of the standard treatment of LD SCLC as the rate of developing brain metastases is very high and PCI has shown to increase overall survival. PCI is given to patients presenting a good response to CHT and tRT. However the overall 5-year rate of brain metastasis with PCI is still very high.

As long as safety data are lacking on PCI administered concurrently with CHT and tRT, PCI is given after the end of CHT in the clinical practice. Therefore the aim of this phase II trial is to evaluate to what extent early HA-PCI given concomitant to CHT and tRT impairs NCF and whether this neurotoxicity can be considered acceptable to evaluate this question in a phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cytologically or histologically confirmed diagnosis of SCLC within 6 weeks before registration.
* Proven LD SCLC (CT thorax, abdomen, and bone scan (or PET/CT only) and brain MRI within 6 weeks before registration) according to the TNM classification version 7 that can be encompassed within a radical radiation port
* Only patients assessed by an interdisciplinary tumor board should be declared eligible taking into account eligibility for curative tRT and CHT according to NCCN Guidelines version 2.2014
* Karnofsky Index ≥ 60%
* Age at registration 18 to 75 years
* Normal bone marrow function: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Calculated creatinine clearance ≥ 60 mL/min is required if chemotherapy with cisplatin is scheduled. If cisplatin has to be replaced by carboplatin a creatinine clearance ≥ 50 mL/min is required
* Normal liver function: bilirubin ≤ 1 x ULN, AST and ALT ≤1.5 x ULN
* Fluency in either German, French or Italian
* Women are not breastfeeding. Women with child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during the 6 months thereafter. A negative pregnancy test before inclusion (within 7 days) into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and during 6 months thereafter.
* Baseline QoL questionnaires FACT-Br and GHQ-12 have been completed within 14 days before registration
* Baseline NCF assessments have been completed within 14 days before registration:

  * HVLT-R
  * COWAT
  * TMT A
  * TMT B
* Patient must give written informed consent before registration

Exclusion Criteria:

* Previous malignancy within 5 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* History of CNS metastases
* Prior brain RT
* History of RT to the thorax
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out QoL forms, participating in assessing NCF testing or interfering with compliance for oral drug intake.
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to trial entry.
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes).
* Any concomitant drugs contraindicated for use with the treatment drugs according to the approved product information.
* History of cerebrovascular disease or epilepsy requiring continuous treatment
* Symptomatic cardiac disease or a history of myocardial infarction within the previous 3 months
* Any psychological, familial or sociological/geographical conditions potentially hampering compliance with the study protocol and follow-up schedule
* Legal incapacity or limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07-11 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Neurocognitive functioning (NCF) | at 6 months
  NCF at 6 months after end of HA-PCI treatment measured by Hopkins Verbal Learning Test Revised (HVLT-R), Controlled Oral Word Association (COWAT) and Trail Making Test Part A and B (TMT A/B). A neurocognitive decline is defined as a decrease of one standard error of measurement (SEM) in any of the four NCF tests.

SECONDARY OUTCOMES:
Brain metastasis free survival (BMFS) | At 6 months and 12 months.
Adverse events according to NCI CTCAE version 4.0 | Until 1 year after the end of HA-PCI treatment.
Neurotoxicity | Until 1 year after HA-PCI treatment.
  Neurotoxicity according to NCI CTCAE version 4.0
Individual tests for each cognitive domain (memory, verbal fluency, visual motor speed, executive function). | At 6 weeks, 6 and 12 months after the end of HA-PCI treatment.
Overall survival (OS) | From time of registration (expected average of 20 months)
Quality of Life (QoL) measured by functional assessment of cancer therapy-brain (FACT-Br) and general health questionnaire (GHQ-12) | At 6 weeks, 6 and 12 months after the end of HA-PCI treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Caparrotti, MD, Study Chair — Hôpitaux Universitaires de Genève, Genève
Locations (8):
- Switzerland (8):
  - Universitätsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopital Fribourgeois, Fribourg
  - Hopitaux Universitaires de Geneve, Geneva
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No